CLINICAL TRIAL: NCT06915454
Title: High-resolution Specimen PET-CT Imaging for the Intraoperative Visualization of Resection Margins: an Exploratory Study
Brief Title: High-Resolution PET-CT Imaging for Surgical Margin Visualization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Vanderbilt University Medical Center (Other); XEOS Medical (Industry)
Responsible Party: Principal Investigator, Michael Topf, Assistant Professor - Head & Neck Surgical Oncology-Microvascular Reconstruction, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCHNP24616
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Solid Malignant Tumors; SCC - Squamous Cell Carcinoma; HNSCC; HNSCC,Larynx, Pharynx and Oral Cavity
Keywords: undergoing surgery; Xeos; PET/CT imaging; specimen scanner; cancer margins; oral cancer; mouth cancer; tongue cancer; gum cancer; scc; head and neck cancer; pharynx; hnscc
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases; Mouth Neoplasms; Tongue Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 18F-FDG (Experimental): After confirming inclusion/exclusion criteria, all participants will receive a one-time IV infusion of 18 F-FDG dose prior to surgical extirpation of tumor. Administration of 18 F-FDG will be injected as a bolus during surgery. Appropriate medical resources for the treatment of severe infusion reactions should be available during infusions, although these are not expected.
  Once the tumor or cancer is resected, it will then be imaged with the XEOS Aura 10 PET/CT Imaging Device.
  Interventions: Device: Intra-op PET/CT Specimen Scanner

INTERVENTIONS:
Device: Intra-op PET/CT Specimen Scanner — Once the tumor or cancer is resected, it will then be imaged with the XEOS Aura 10 PET/CT Imaging Device. Imaging will be obtained utilizing a XEOS AURA 10 scanner in real time while in the operating room with the surgery team still present.
  Other Names: XEOS Aura 10

SUMMARY:
Imaging will be exploratory and be used intraoperatively. There have been no discovered risks associated with the device to be used in this study, and none are anticipated given the diagnostic and non-invasive, 'ex vivo' nature of device use. Of note, the surgical resection will proceed as per standard of care and will not be affected by the research protocol.

Potential Benefit: Imaging intra-operatively will ensure surgeons to identify at risk resection margins.

Time Commitment: There are no additional visits that will be asked of you to partake in this study.

Drug is FDA approved and Exposure to Radiation is minimal.

DETAILED DESCRIPTION:
This pilot study explores the use of high-resolution PET imaging to identify surgical margins in solid tumors after removal. It evaluates the feasibility and potential of using PET-CT to assess tumor specimens and ensures radiation safety with a low-dose 18-FDG injection (20% of the standard dose). Previous studies have shown good tumor visualization in breast, pancreatic, prostate, and head and neck tumors, supporting the method's proof-of-concept. This research aims to gather insights into its clinical usefulness across different cases

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of any solid malignancy
* Diagnosis of any T stage, any subsite that are scheduled to undergo definitive en bloc surgical resection. Patients with recurrent disease or a new primary will be allowed.
* Planned standard of care oncologic surgery with curative intent
* Male or female patients age ≥ 18 years
* Have life expectancy of more than 12 weeks
* Karnofsky performance status of at least 70% or ECOG/Zubrod level 1
* Have acceptable glucose status (<200 mg/dL) at Day of Surgery prior to 18F-FDG injection

Exclusion Criteria:

* General or local contraindications for resective surgery
* Women who are pregnant or breast-feeding
* Blood glucose level over 200 mg/dL prior to 18F-FDG infusion
* Any participation in other clinical trials or research study that involved a radiation exposure of more than 1 mSv in the past year. If the participant had radiation exposure greater than 1 mSv as SOC, they would not be excluded unless the Principal Investigator determines that patient could be at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The study will determine the feasibility of intraoperative high-resolution specimen PET-CT imaging in solid tumors. | Day of Surgery.
  This study is an exploratory pilot study where the main goal is to gather scientific knowledge. Since no results with a certain significance need to be proven, no power analysis will be performed.
  Pre-Surgery Preparation: Patients are injected with a PET (18F-FDG) tracer. This tracer highlights cancerous tissues by emitting signals detectable by PET imaging.
  Intraoperative Imaging: Once the tumor is removed, the specimen is scanned using the XEOS Aura 10 device in the operating room. This allows surgeons to get detailed images of the tumor and surrounding tissues.
  Immediate Analysis: The imaging provides real-time feedback on the tumor's characteristics, such as margins and whether all cancerous tissue has been removed. This can help surgeons make decisions during the operation, like whether additional tissue needs to be excised.
  Comparison with Pathology: The PET-CT images are later compared with traditional pathology results to validate their accuracy and usefulness.

SECONDARY OUTCOMES:
Correlate the margin status based on high-resolution specimen PET-CT images with the actual margin status based on gold standard microscopic histopathological analysis; | Day of Surgery to Pathology
  Researchers will compare pathology data that is to be completed as standard of care to the XEOS Aura 10 specimen scanner margins.
Correlate lymph node status based on high-resolution specimen PET-CT images with the actual lymph node status based on gold standard microscopic histopathological analysis | Day of Surgery to Pathology
  Researchers will compare pathology data that is to be completed as standard of care to the XEOS Aura 10 specimen scanner margins.
Compare the visualization of the target lesion between intraoperative high-resolution specimen PET-CT imaging and pre-operative whole-body PET-CT imaging (when performed per standard of care oncologic work-up). | Day of Surgery to 10 days.
  Researchers will compare standard of care imaging data to the XEOS Aura 10 specimen scanner data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Topf, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the data and key findings from our pilot study, which explored the feasibility and potential of high-resolution PET imaging for assessing surgical margins in solid tumors. This information will be made available to support further research, foster collaboration, and provide insights into the clinical application of ex vivo PET-CT imaging in oncology. Our findings include promising results from studies on various tumor types, highlighting the technique's ability to visualize tumors effectively with a low-dose radiation protocol.

DOCUMENTS (1):
  • Informed Consent Form (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT06915454/ICF_000.pdf